CLINICAL TRIAL: NCT03609333
Title: Characterizing the cerebrovAscular Physiology of Optimal Mean Arterial Pressure Targeted Resuscitation in Hypoxic Ischemic Brain Injury After Cardiac Arrest
Brief Title: Characterizing the cerebrovAscular Physiology of Optimal Mean Arterial Pressure Targeted Resuscitation
Acronym: CAMPHIBIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Myp Sekhon, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Purpose: Basic Science
Other Study IDs: H16-00466
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internal arm (Experimental)
  Interventions: Device: Multimodal Neuromonitoring

INTERVENTIONS:
Device: Multimodal Neuromonitoring — Application of multimodal neuromonitoring
  Other Names: Targeted optimal MAP resuscitation

SUMMARY:
Hypoxic ischemic brain injury is a devastating illness that occurs after cardiac arrest (the heart stopping) and can yield irreversible brain damage, often leading to death. The mainstay in therapy is to optimize the delivery of oxygen to the brain to help it recover. In patients with traumatic brain injury (similar to HIBI), the investigators are able to optimize oxygen delivery to the brain with the use of wires placed into the brain that sense the pressure and oxygen in the skull to find the ideal blood pressure for each individual patient. This strategy is associated with improved outcomes. The investigators are conducting a prospective study investigating whether the perfusion within proximity to the optimal MAP is associated with improved brain oxygenation and blood flow .

ELIGIBILITY:
Inclusion Criteria:

* Confirmed cardiac arrest with return of spontaneous circulation > 10 minutes
* post resuscitation GCS < 9

Exclusion Criteria:

* concurrent coagulopathy
* prior history of TBI, intracranial hemorrhage, subarachnoid hemorrhage
* anticipated cardiac catheterization within next 7 days
* anticipated or current use of anticoagulants or anit-platelets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11-12 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Cerberal blood flow | 12 hours
  mls/100g/min

CONTACTS AND LOCATIONS:
Overall Officials: Mypinder Sekhon, MD, Principal Investigator — UBC
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sekhon MS, Ainslie PN, Menon DK, Thiara SS, Cardim D, Gupta AK, Hoiland RL, Gooderham P, Griesdale DE. Brain Hypoxia Secondary to Diffusion Limitation in Hypoxic Ischemic Brain Injury Postcardiac Arrest. Crit Care Med. 2020 Mar;48(3):378-384. doi: 10.1097/CCM.0000000000004138. PMID 31789834
- [Derived] Sekhon MS, Griesdale DE, Ainslie PN, Gooderham P, Foster D, Czosnyka M, Robba C, Cardim D. Intracranial pressure and compliance in hypoxic ischemic brain injury patients after cardiac arrest. Resuscitation. 2019 Aug;141:96-103. doi: 10.1016/j.resuscitation.2019.05.036. Epub 2019 Jun 8. PMID 31185256